CLINICAL TRIAL: NCT05139134
Title: Immunohistochemical Expression of CXCL5 as a Valuable Prognostic Marker in Urinary Bladder Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-21-10-43
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Urinary Bladder Urothelial Carcinoma
Keywords: CXCL5; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urothelial carcinoma is common malignant tumor worldwide, it remains a challenge in the oncology field, it is an ideal for research on biomarkers that could identify tumor progression and prognosis. CXCL5 have been implicated in progression of many cancers, but their significance in urinary bladder UC remains unclear.

DETAILED DESCRIPTION:
Bladder carcinoma has become a common cancer globally, Incidence rates are highest in Europe, the United States and Egypt. In Egypt, bladder carcinoma was considered the third most common tumor; Egyptian males have the highest mortality rates. UC of the urinary bladder represents about 90% of all bladder cancers.

CXCL5 is a chemokine, belonging to ‗ELR+' subgroup. It plays an important role in angiogenesis and tumor migration. Numerous reports have indicated that CXCL5 plays important roles in cancer progression, including cholangiocarcinoma, prostate cancer, and gastric cancer. Studying the IHC expression of CXCL5 in UC to assess its role in tumor cell proliferation, migration and spread is needed.

ELIGIBILITY:
Inclusion Criteria:Patients with primary invasive and non-invasive urinary bladder urothelial carcinomas.

-

Exclusion Criteria:

* - Patients received pre-operative chemotherapy or radiotherapy.
* Patients with insufficient clinical data.
* Specimens with extensive necrosis
* Tiny specimens which are insufficient for accurate diagnosis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Fifty specimens of urothelial carcinoma obtained from patients in Urology Department of Sohag Faculty of Medicine,
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
assess the expression of CXCL5 in urothelial carcinoma | 1 month
  Immunohistochemical study

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ahmed, Lecturer, Principal Investigator — Sohag University
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt